CLINICAL TRIAL: NCT03952936
Title: Vestibular Rehabilitation for Chronic Central Vestibular Deficits Due to Cerebellar Dysfunction
Brief Title: Vestibular Rehabilitation for Chronic Central Vestibular Deficits: A Case Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Methodist University, North Carolina (Other)
Responsible Party: Principal Investigator, Stacia Hall, Assistant Professor of Physical Therapy, Methodist University, North Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5/14/2020 CVD
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Vestibular Disorder; Fall; Coordination and Balance Disturbances
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Intervention Model Description: Case study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobility (Other): Self comparison of data from pre-post intervention.
  Interventions: Other: Vestibular Rehabilitation

INTERVENTIONS:
Other: Vestibular Rehabilitation — standard vestibular rehabilitation with gaze stability, balance training, habituation tailored to the subject

SUMMARY:
The purpose of this study is to assess the effectiveness of vestibular rehabilitation for an individual who has chronic central vestibular deficits due to cerebellar dysfunction. Due to the lack of treatment for chronic cerebellar dysfunction with Physical Therapy, the investigators hope to produce a protocol for chronic cerebellar dysfunction utilizing balance training, vestibular rehabilitation, or any other rehabilitation technique that may alleviate or eliminate symptoms.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effectiveness of vestibular rehabilitation for an individual who has chronic central vestibular deficits due to cerebellar dysfunction. Due to the lack of treatment for chronic cerebellar dysfunction with Physical Therapy, the investigators hope to produce a protocol for chronic cerebellar dysfunction utilizing balance training, vestibular rehabilitation, or any other rehabilitation technique that may alleviate or eliminate symptoms.

Investigators will test the subject initially at 4 weeks, 8 weeks and 6 months post start date to assess for symptom improvement.

ELIGIBILITY:
Inclusion Criteria:

* Central vestibular deficits

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Activity Specific Balance Confidence Scale | 2-6 months
  Perceived self confidence with balance. 16 items are scored on a 0-100% scale. Items are totaled and then averaged. The higher the average score the higher the confidence with balance and the less likely risk there is for falling.

SECONDARY OUTCOMES:
Dizziness handicap inventory | 2-6 months
  Perceived handicap from dizziness. Items are scored on a 0, 2 or 4 point scale with adding up the total number of the 26 items. The lower the score, the less perceived amount of handicap is present.
Functional Gait Assessment | 2-6 months
  Gait and balance test. 10 item test rated on each item from 0-3. total score is calculated of 10 items. the higher the score the less likely risk for falling is present.
Motion Sensitivity Quotient | 2-6 months
  Motion sickness indicator. 16 items are scored based on symptom severity and duration. positive items are calculated together to receive a percentage. the lower the percentage the less motion sensitivity a person has.
Modified Clinical Test for Sensory Integration in Balance | 2-6 months
  balance test for sensory system inputs. 6 item test to check for sensory integration with balance. each of the 6 items is calculated for length of time and amount of sway. the less the sway, the lower the score and the better the balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Methodist Universtiy, Fayetteville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No